CLINICAL TRIAL: NCT05492071
Title: Vibration Mediated Dilation and Flow Mediated Dilation in Human Circulatory System
Brief Title: Impact of Regional Vibration Application and Flow Mediated Dilation on Brachial Artery Hemodynamics
Acronym: VMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr. Murat Sezer, Professor, MD, Istanbul University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020/755
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Vasodilation; Diabetes Mellitus, Type 2
Keywords: Vibration; Peripheral Artery Hemodynamics; Diabetes Mellitus
MeSH Terms: conditions — Aneurysm; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local Vibration Application Following Flow-Mediated Dilation Application (Experimental): Flow mediated dilatation will be induced via 5 min cuff inflation below left elbow at suprasystolic pressures (50mmHg above preapplication systolic pressure). Vibration is applied with a commercially available vibration plate to forearm at 20 hz and 3 mm of vertical amplitude for 5 minutes, 30 minutes after termination of FMD.
  Interventions: Device: Local Vibration Application Following Flow Mediated Dilation
- Flow-Mediated Dilation Application (Experimental): Flow mediated dilatation will be induced via 5 min cuff inflation below left elbow at suprasystolic pressures (50mmHg above preapplication systolic pressure).
  Interventions: Other: Flow mediated dilation

INTERVENTIONS:
Device: Local Vibration Application Following Flow Mediated Dilation — Flow mediated dilatation will be induced via 5 min cuff inflation below left elbow at suprasystolic pressures (50mmHg above preapplication systolic pressure). Vibration is applied with a commercially available vibration plate to forearm at 20 hz and 3 mm of vertical amplitude for 5 minutes, 30 minutes after termination of FMD.
  Arms: Local Vibration Application Following Flow-Mediated Dilation Application
Other: Flow mediated dilation — Flow mediated dilatation will be induced via 5 min cuff inflation below left elbow at suprasystolic pressures (50mmHg above preapplication systolic pressure).
  Arms: Flow-Mediated Dilation Application

SUMMARY:
Application of vibration has been previously shown to affect tissue perfusion and utilized in different branches of medicine. Little is known about the acute impact of vibration application on peripheral artery hemodynamics. In this study, investigators intend to assess:

1. vibration induced hemodynamic changes in brachial artery in non-diabetic patients and compare the characteristics of these alterations with flow mediated dilation mediated changes in same cohort.
2. compare the characteristics of vibration mediated hemodynamic alterations in diabetic and non-diabetic subgroups.

DETAILED DESCRIPTION:
Background and Rationale:

Vibration application has been previously shown to affect tissue perfusion and utilized in different branches of medicine. However, previous studies have mainly focused on the impact of vibration on skin perfusion or vibration with active muscle contractions, therefore couldn't truly demonstrate acute impact of local vibration application on peripheral arteries. In addition to that, as a population that is prone to develop vascular problems, it is not known whether diabetic patients have comparable response to vibration application with non-diabetic population.

Objectives:

In this study, investigators aim to demonstrate and compare hemodynamic alterations in brachial artery with paired measurements pre- and post- vibration application and compare the characteristics of these changes with those of flow-mediated dilation in a non-diabetic cohort. Additionally, differences and similarities in vascular hemodynamic response to vibration in diabetic and non-diabetic subgroups are intended to be elucidated.

Methods:

Flow mediated dilatation and vibration will be applied after the participants will abstain from alcohol, caffeine and nicotine for 24 hours. Flow mediated dilatation (FMD) will be induced via 5 min cuff inflation below left elbow at supra-systolic pressures (50mmHg above pre-application systolic pressure). Vibration will be applied with a commercially available vibration plate to forearm at 20 hz and 3 mm of vertical amplitude for 5 minutes, 30 minutes after termination of FMD. Left Brachial artery flow will be measured with pulsed Doppler and diameter will be measured via 2D ultrasonographic imaging at 0th, 2nd, 4th, 6th, 8th minutes.Throughout the entire application and measurement periods, patients will be continuously monitored with electrocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 80
* Sinus Rhythm in ECG
* Ejection Fraction > %35
* Informed Consent

Exclusion Criteria:

* Unstabile angina
* Certain or suspected subclavian artery or brachial artery atherosclerotic disease (assessed with USG)
* Heart failure ( New York Heart Association III - IV)
* Atrial fibrillation or frequent extrasystoles in ECG.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Brachial Artery Diameter | Up to 10 minutes after vibration application initiation
  vessel diameter in millimeters
Brachial Artery Mean Flow Velocity | Up to 10 minutes after vibration application initiation
  Mean flow velocity ( cm/sec) measured with Doppler

OTHER OUTCOMES:
Magnitude of Maximum Blood Flow Change | Up to 10 minutes after vibration application initiation
  Magnitude of Maximum Blood Flow Change in Diabetic and Nondiabetic subgroups
Magnitude of Maximum Diameter Change | Up to 10 minutes after vibration application initiation
  Magnitude of Maximum Diameter Change in Diabetic and Nondiabetic subgroups
Magnitude of Maximum Resistance Change | Up to 10 minutes after vibration application initiation
  Magnitude of Maximum Resistance Change in Diabetic and Nondiabetic subgroups
Magnitude of Maximum Mean Flow Velocity Change | Up to 10 minutes after vibration application initiation
  Magnitude of Maximum Mean Flow Velocity Change in Diabetic and Nondiabetic subgroups

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Department of Cardiology, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Herrero AJ, Menendez H, Gil L, Martin J, Martin T, Garcia-Lopez D, Gil-Agudo A, Marin PJ. Effects of whole-body vibration on blood flow and neuromuscular activity in spinal cord injury. Spinal Cord. 2011 Apr;49(4):554-9. doi: 10.1038/sc.2010.151. Epub 2010 Nov 2. PMID 21042329
- [Background] Robbins D, Yoganathan P, Goss-Sampson M. The influence of whole body vibration on the central and peripheral cardiovascular system. Clin Physiol Funct Imaging. 2014 Sep;34(5):364-9. doi: 10.1111/cpf.12103. Epub 2013 Nov 17. PMID 24237890
- [Background] Aoyama A, Yamaoka-Tojo M, Obara S, Shimizu E, Fujiyoshi K, Noda C, Matsunaga A, Ako J. Acute Effects of Whole-Body Vibration Training on Endothelial Function and Cardiovascular Response in Elderly Patients with Cardiovascular Disease. Int Heart J. 2019 Jul 27;60(4):854-861. doi: 10.1536/ihj.18-592. Epub 2019 Jun 28. PMID 31257335